CLINICAL TRIAL: NCT00659217
Title: Effect of Mesenchymal Stem Cell Transplantation for Lupus Nephritis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Organ Transplant Institute, China (Other Government)
Responsible Party: FUZHOU GENERAL HOSPITAL, FUZHOU GENERAL HOSPITAL
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: fuzhough0713
Record Dates: First submitted 2008-04-14; First posted 2008-04-16 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2008-04

CONDITIONS: Lupus Nephritis
Keywords: Mesenchymal Stem Cells; lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 (Experimental): mesenchymal stem cell Autologous MSC transplantation
  Interventions: Biological: mesenchymal stem cell

INTERVENTIONS:
Biological: mesenchymal stem cell — Autologous MSC transplantation

SUMMARY:
Mesenchymal Stem Cell (MSC) has been shown to have immunosuppressive and repairing properties. Manifestations of systemic lupus eryhematosus(SLE) may in most patients be ameliorated with medications that suppress the immune system. Nevertheless, there remains a subset of SLE patients for whom current strategies are insufficient to control disease. The investigators will infuse expanded autologous MSC into patients with lupus Nephritis. The purpose of this trial is to evaluate whether this new therapeutical approach will result in improvement in the lupus disease.

DETAILED DESCRIPTION:
Mesenchymal stem cells (MSC), or marrow stromal cells, are multipotential cells that reside within the bone marrow and can be induced to differentiate into various components of the marrow microenvironment, such as bone, adipose and stromal tissues under proper conditions. It has been reported that MSCs can suppress maturation, activation and proliferation of T, B, NK and DC cell in vitro and downregulate immune response in vivo. MSCs are presently being cotransplantated with hematopoietic stem cell, which can facilitates engraftment of hematopoietic stem cells and prevent GVHD. Systemic lupus erythematosus (SLE) is an autoimmune disorder that affects many organ systems. Autoimmune diseases are illnesses that occur when the body's tissues are attacked by its own immune system. Patients with lupus produce abnormal antibodies in their blood that target tissues within their own body. Because the antibodies and accompanying cells of inflammation can involve tissues anywhere in the body, lupus has the potential to affect a variety of areas of the body. The origin of autoantibody production in SLE is unclear but a role has been suggested for an antigen driven process, spontaneous B-cell hyper-responsiveness, or impaired immune regulation.

The BXSB mouse strain spontaneously develops a progressive and lethal autoimmune disease, similar to human SLE. In our previous work we found that transplantation of MSCs could alleviate the symptoms of BXSB mouse.

This study will evaluate the safety and effectiveness of expanded autologous MSC infusions in patients with primary and treatment -refractory SLE. This study will last 2 years. Participants will be assigned to receive either the prednisone (Group 1) or MSC infusions alone (Group 2). Patients will undergo MSC infusions at the start of the study on Day 0. One year post- infusions, Patients will be clinically assessed and evaluated for MSC and disease response, and participants will undergo kidney biopsies at 12 Months.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 to 50 years old.
2. Meet at least 4 of 11 American College of Rheumatology (ACR) Classification criteria for SLE.
3. Able to give informed consent.
4. For treatment -refractory lupus nephritis, participants must fail pulse cyclophosphamide, a renal biopsy must be obtained and document either class III or IV glomerulonephritis.

Exclusion Criteria:

1. Pregnant women.
2. Previous history of malignancy
3. Active infection including hepatitis B, hepatitis C, HIV, or TB as determined by a positive skin test or clinical presentation, or under treatment for suspected TB.
4. Evidence of cardiovascular disease, existing congestive cardiac failure on physical exam and/or acute coronary syndrome in past 6 months.
5. Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible.
6. Transaminases greater than 2 times normal unless due to active lupus.
7. Any illness that in the opinion of the investigator would jeopardize the ability of the Patient to tolerate this treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
the proportion of participants who achieve and maintain remission | 5

SECONDARY OUTCOMES:
Patient survival | 5
Creatinine and proteinuria. | 5
SLE disease activity index | 5
Serology (ANA, dsDNA) | 5
ComplementC3 and C4 | 5

CONTACTS AND LOCATIONS:
Locations (1):
- Fuzhou General Hospital, Fuzhou, Fujian, China